CLINICAL TRIAL: NCT03088111
Title: A Phase 4, Open Label Field Study to Evaluate the Clinical Benefit, Safety, and Pharmacokinetics of Anthim (Obiltoxaximab) When Used in the Treatment of Suspected, Probable, or Confirmed Cases of Inhalational Anthrax Due to B. Anthracis
Brief Title: An Open Label Field Study of Anthim (Obiltoxaximab) in Subjects Exposed to B. Anthracis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Elusys Therapeutics (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); APCER Life Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AH501; HHSO100201100034C (Other Grant/Funding Number: Biomedical Advanced Research and Development Authority)
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Infection, Bacterial; Anthrax
Keywords: Anthim®; Obiltoxaximab; anthrax; anti-toxin
MeSH Terms: conditions — Bacterial Infections; Anthrax | interventions — obiltoxaximab

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Obiltoxaximab (Other): This is an open label, 24-week, single arm field study that will be implemented for subjects who receive FDA-approved obiltoxaximab as part of their medical treatment for inhalational anthrax infection in the United States. Adult subjects will be administered a single, intravenous (IV) dose of 16 mg/kg obiltoxaximab given as part of their medical care. Children will receive a weight-adjusted dose.
  The primary purpose of the study is to collect data from subjects who have been treated with obiltoxaximab as part of their medical care for inhalational anthrax and to collect additional blood samples for measurement of obiltoxaximab concentrations and presence of anti-therapeutic antibodies (ATA).
  Interventions: Other: Collection of samples; Biological: Obiltoxaximab

INTERVENTIONS:
Other: Collection of samples — To the extent possible, blood samples will be collected from all subjects prior to infusion and at specified time points post-infusion to determine serum obiltoxaximab concentrations and ATA titers. Scavenged blood samples can be utilized, if acceptable, to maximize sample analyses for pharmacokinetic and other investigational parameters. Data on other relevant laboratory testing will only be collected and evaluated if available in the subject's record (eg, protective antigen (PA), anti-PA, anti-lethal factor (LF), anti-edema factor, IgG antibodies, anthrax lethal toxin neutralizing activity, presence of anthrax LF, incidence and duration of B. anthracis bacteremia, and demonstration of B. anthracis antigens in tissues).
Biological: Obiltoxaximab — Obiltoxaximab standard of care
  Other Names: Anthim

SUMMARY:
This field study is a post-marketing requirement from the FDA to evaluate the clinical benefit (course of illness and survival), safety and pharmacokinetics of obiltoxaximab administered to patients as part of their medical care for treatment or prophylaxis of inhalational anthrax infection following exposure to Bacillus anthracis (B. anthracis). The protocol can be implemented for any individual who receives obiltoxaximab for a suspected, probable, or confirmed case of inhalational anthrax due to B. anthracis in the United States, including sporadic cases, small incidents and/or a mass event. In case of a small anthrax incident, to the extent possible, the information will be collected prospectively at prespecified time points, except where it would interfere with management of the subject's illness. However, because of the logistical complexities that would likely accompany a mass anthrax event, most data in this study are anticipated to be collected retrospectively. Both retrospective and prospective data collection are allowed to maximize information collection. This study will collect data on the use of obiltoxaximab in anthrax infected or exposed subjects and the data collected will inform the understanding of the clinical benefit and safety of obiltoxaximab.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (including pregnant and lactating women) and children of all ages who receive obiltoxaximab as part of their clinical care for anthrax infection and are willing and able to give written informed consent themselves or through legally acceptable representative (for minors, unconscious adults or deceased subjects) to participate in the study

Exclusion Criteria:

* There are no exclusion criteria defined for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival in suspected, probable, or confirmed cases of inhalational anthrax at Week 24 | Up to Week 24
  Overall survival will be summarized by frequency of subjects who completed the study at Week 24, and subjects who died before that visit. Population survival distribution function (SDF) will be estimated using the Kaplan-Meier (KM) method.

SECONDARY OUTCOMES:
Survival at Day 14 and Day 28 | Up to Day 28
  Population survival rates at 14 and 28 days will be estimated using the KM method.
Duration of survival (to Week 24) | Up to Week 24
  The KM method will be used to estimate duration of survival.
Disease progression and associated complications rates of anthrax (meningitis, pleural effusion, ventilator support) (to Week 24) | Up to Week 24
  The progression to systemic anthrax infection and complication rates will be summarized using KM estimates associated with time to disease progression and time to complication of anthrax. The population SDFs of time to progression to systemic anthrax infection and of time to complication will be estimated using the KM method. Summary statistics of subjects with disease progression and complication rates will be provided.
Modified SOFA score (to Week 24) | Up to Week 24
  Modified sequential organ failure assessment (SOFA) scores will be assessed using 5 organ systems (respiratory, liver, cardiovascular, central nervous system, renal).
Incidence and duration of B. anthracis bacteremia | Up to Week 24
  Incidence and duration of B. anthracis bacteremia will be summarized by total incidence across time points of subjects with bacteremia and time from study drug administration to onset of bacteremia.

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Clinical Development, Study Director — NightHawk Biosciences; Timothy S. Leach, MD, MPH, Study Director — Contract Medical Monitor

IPD SHARING:
Plan to Share IPD: Undecided